CLINICAL TRIAL: NCT02241772
Title: A Study on the Effects of TA-8995 on Lp(a) in Subjects With Elevated Lp(a)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xention Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-8995-06
Record Dates: First submitted 2014-08-20; First posted 2014-09-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2014-10

CONDITIONS: Elevated Lp(a)
MeSH Terms: interventions — TA-8995

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 10mg TA-8995 (Experimental): 10mg TA-8995 once daily
  Interventions: Drug: TA-8995
- 2.5mg TA-8995 (Experimental): 2.5mg TA-8995 once daily
  Interventions: Drug: TA-8995
- Placebo to TA-8995 (Placebo Comparator): Placebo to TA-8995 once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TA-8995
  Arms: 10mg TA-8995; 2.5mg TA-8995
Drug: Placebo
  Arms: Placebo to TA-8995

SUMMARY:
A study in males and females with elevated Lp(a) to look at the effects of TA-8995 on Lp(a) levels.

ELIGIBILITY:
Inclusion Criteria:

* Male and female (of non-child bearing potential) subjects with elevated Lp(a) levels

Exclusion Criteria:

* Clinically significant medical history
* Abnormal laboratory results (other than lipid levels) or vital signs
* Receiving any other drug therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the change from baseline in (Lp(a) levels after 12 weeks of treatment with TA-8995. | 12 weeks

SECONDARY OUTCOMES:
Number of participants with adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev Hospital, Herlev, Denmark